CLINICAL TRIAL: NCT02106741
Title: Randomized Pilot Study of Self-Administered Acupressure for Patients With Low Back Pain
Brief Title: Acupressure for Fatigue and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor, Department of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAK
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2015-08

CONDITIONS: Fatigue; Chronic Low Back Pain
Keywords: Pain; Acupressure; Symptoms; Fatigue; Self-administered
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Relaxation acupressure (Experimental)
  Interventions: Behavioral: Relaxation acupressure
- Stimulating acupressure (Active Comparator)
  Interventions: Behavioral: Stimulating acupressure
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: Relaxation acupressure — The relaxation acupressure protocol will use a set of nine fixed acupoints: forehead, twixt the eyebrows (unilateral); posterior neck, behind the ears (bilateral); palmer side of hand at wrist (bilateral); inside of lower leg (bilateral); top of foot (bilateral).
  A trained acupressure educator will meet with each participant and demonstrate the sites and techniques for self-administered acupressure. Additionally, each participant will receive a demonstration DVD and a laminated handout detailing the locations of each acupoint.
  Participants will be asked to perform daily acupressure sessions using the assigned sites. Each site is stimulated for 3 minutes, and the entire session can be completed in approximately 30 minutes.
  Arms: Relaxation acupressure
Behavioral: Stimulating acupressure — The stimulating acupressure protocol will use a set of ten fixed acupoints: top of the head (unilateral); below the navel (unilateral); back of the hand (bilateral); outside of lower leg (bilateral); inside of lower leg (bilateral); inside of ankle (bilateral).
  A trained acupressure educator will meet with each participant and demonstrate the sites and techniques for self-administered acupressure. Additionally, each participant will receive a demonstration DVD and a laminated handout detailing the locations of each acupoint.
  Participants will be asked to perform daily acupressure sessions using the assigned sites. Each site is stimulated for 3 minutes, and the entire session can be completed in approximately 30 minutes.
  Arms: Stimulating acupressure

SUMMARY:
The purpose of this study is to compare two kinds of self-administered acupressure (relaxation acupressure and stimulating acupressure) to usual care for management of fatigue and pain in low back pain patients.

Hypothesis: Self-administered relaxation acupressure will result in improvements in fatigue and sleep quality, pain, and physical function compared to stimulating acupressure and usual care.

DETAILED DESCRIPTION:
Acupressure is a Traditional Chinese Medicine (TCM) technique based on a philosophy similar to that of acupuncture. It involves the application of physical pressure on different acupuncture points (acupoints). One advantage of acupressure is the ability to self-administer the treatment. Acupressure is also a viable alternative to acupuncture in situations where patients: (1) cannot come to the clinic to receive an acupuncture treatment; (2) when a more frequent intervention is needed; or (3) where needle phobia or safety concerns are an issue.

The objective of this study is to evaluate the validity and feasibility of teaching acupressure interventions using an acupressure educator for the management of symptoms related to low back pain.

Specific aims:

1. To examine the effect of 6-weeks of relaxation acupressure (RA) compared to a regime of stimulating acupressure (SA) or wait-list control (WL) on fatigue and sleep quality as assessed by Brief Fatigue Inventory and wrist-worn accelerometry (sleep efficiency).
2. To explore the effect of 6-weeks of RA compared to a regime of SA or WL on for chronic low back pain in terms of reduced pain and improved function.

ELIGIBILITY:
Inclusion Criteria:

* Aged18-65 years
* Non-specific low back pain (either by self-report or via ICD-9 codes 724.2, 724.5, 846.0-846.9)
* Low back pain that has persisted for at least 3 months
* Minimum of 3/10 on the Pain Bothersome Scale
* Minimum of 3/10 fatigue severity
* Ambulatory with or without assistive device
* Ability to operate the accelerometer (Actiwatch-S)
* Stable medication regiment for the previous 2 months
* Report of a physician's visit during the previous 24 months
* English-speaking

Exclusion Criteria:

* Medically unstable (acute conditions or acute presentations of chronic conditions)
* Current pregnancy
* Radiculopathy or report of low back pain radiating to below the knee
* Reported history of spinal fracture, herniated lumbar disc, ankylosing spondylitis, and spinal stenosis.
* Report of back surgery within the preceding 12 months
* Participation in active litigation or compensation claims
* Conditions that might confound treatment effects or interpretation of results (for example, rheumatoid arthritis, lupus)
* Acupuncture or acupressure within the preceding 12 months
* Report of sleep apnea
* 2nd or 3rd shift workers or other non-traditional sleep schedules
* Use of anti-coagulant/platelet therapy within the preceding month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Fatigue severity and interference in daily activities | Week 0 (baseline) and approximately 9 weeks (follow-up)
  Fatigue severity and interference in daily activities will be measured using the Brief Fatigue Inventory. Subjects will answer the BFI at both baseline and follow-up. To investigate a change from baseline in fatigue, the difference between the post-assessment outcomes and baseline measures will be calculated. Analyses on these differences will be performed using independent samples t-tests between treatment groups. We will also evaluate all continuous outcomes by ANCOVA, adjusting for baseline value and treatment group.
Sleep quality via objectively measured sleep efficiency | Week 0 (baseline) and approximately 9 weeks (follow-up)
  We will use wrist-worn accelerometry to assess sleep efficiency. Subjects will wear a wrist-worn accelerometer for 7 consecutive days (at baseline and follow-up) that collects in vivo sleep quality data; an accompanying logbook will be used to enhance objective data. To investigate a change from baseline in sleep efficiency, the difference between the post-assessment outcomes and baseline measures will be calculated. Analyses on these differences will be performed using independent samples t-tests between treatment groups. We will also evaluate all continuous outcomes by ANCOVA, adjusting for baseline value and treatment group.

SECONDARY OUTCOMES:
Pain severity and interference in daily activities | Week 0 (baseline) and approximately 9 weeks (follow-up)
  Pain severity and interference in daily activities will be measured using the Brief Pain Inventory. Subjects will answer the BPI at both baseline and follow-up. To investigate a change from baseline in pain, the difference between the post-assessment outcomes and baseline measures will be calculated. Analyses on these differences will be performed using independent samples t-tests between treatment groups. We will also evaluate all continuous outcomes by ANCOVA, adjusting for baseline value and treatment group.
Level of physical functioning as measured by the Roland-Morris Disability Questionnaire. | Week 0 (baseline) and approximately 9 weeks (follow-up)
  Subjects will answer the Roland-Morris Disability Questionnaire at both baseline and follow-up. To investigate a change from baseline in physical function, the difference between the post-assessment outcomes and baseline measures will be calculated. Analyses on these differences will be performed using independent samples t-tests between treatment groups. We will also evaluate all continuous outcomes by ANCOVA, adjusting for baseline value and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Murphy, ScD, OTR, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy SL, Harris RE, Keshavarzi NR, Zick SM. Self-Administered Acupressure for Chronic Low Back Pain: A Randomized Controlled Pilot Trial. Pain Med. 2019 Dec 1;20(12):2588-2597. doi: 10.1093/pm/pnz138. PMID 31237610